CLINICAL TRIAL: NCT03116126
Title: Randomised Clinical Trial of Noradrenergic Add-on Therapy With Extended-Release Guanfacine in Alzheimer's Disease
Brief Title: Noradrenergic Add-on Therapy With Guanfacine
Acronym: NorAD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRAS 171996
Record Dates: First submitted 2017-04-04; First posted 2017-04-14 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guanfacine (Active Comparator)
  Interventions: Drug: Guanfacine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine — 2mg oral daily tablet
  Arms: Guanfacine
Drug: Placebo — inactive oral daily tablet
  Arms: Placebo

SUMMARY:
NorAD is a clinical trial funded by the UK National Institute of Health Research. In this trial the investigators will assess whether a long-acting preparation of guanfacine, a drug used to treat Attention Deficit Hyperactivity Disorder in children, can improve thinking (particularly attention) in Alzheimer's Disease when it is added to the standard NICE-approved drugs that are normally used in this condition.

This is a randomized clinical trial designed to evaluate the efficacy of extended-release guanfacine as an add-on therapy in AD, and whether it improves cognition compared to standard cholinergic therapy alone.

DETAILED DESCRIPTION:
There is evidence suggesting that both noradrenaline and acetylcholine have key roles to play in attention. Guanfacine acts by increasing levels of noradrenaline, a substance in the brain which is closely linked with attention, both noradrenaline levels and attentional performance have been shown to be reduced in Alzheimer's Disease.

In this study the investigators propose that modulation of the noradrenergic deficit that has been described in Alzheimer's Disease in addition to standard cholinergic treatment could have significant positive effects on cognition, particularly in those patients who suffer from attentional impairments. The investigators want to assess whether long-acting guanfacine should be used in addition to NICE-approved drugs that are currently being used in AD as part of combination therapy.

It is a single-centre, randomised, parallel-group, double-blind controlled Phase 3 trial to compare the efficacy of standard cholinergic therapy (Donepezil, Rivastigmine or Galantamine) plus extended release guanfacine (2mg GXR) versus standard cholinergic therapy plus placebo on Cognition (as measured by the ADAS-Cog) in patients with mild to moderate Alzheimer's Disease.

The trial, which will recruit 160 patients (80 randomised to GXR add-on therapy and 80 randomised to placebo), based at Imperial College London - Imperial College Healthcare NHS Trust.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* NINCDS/ADRDA criteria for probable AD
* MMSE at assessment = 10-30
* Identified informant to accompany patient at all visits
* Stable dose of donepezil, galantamine or rivastigmine for preceding 12 weeks

Exclusion Criteria:

* Labile blood pressure or new antihypertensive medication started within 3 weeks
* Severe coronary insufficiency or myocardial infarction in previous 6 months
* History of unexplained syncope within the preceding 12 months
* Cardiac Conduction Block
* Severe Hepatic Impairment (ALT > 120 (Upper Limit of Normal (ULN) is 40) OR Alkaline Phosphatase > 390 (ULN 130)) OR Both ALT and total bilirubin > ULN OR Total bilirubin > 60 (ULN 30)
* Severe Renal Impairment (eGFR < 40)
* Treatment with other medications known to potentiate guanfacine's hypotensive effects or cause arrhythmia (specifically antipsychotics (including sultopride, chlorpromazine, thioridazine, amisulpiride, sulpiride, haloperidol), and moxifloxacin, baclofen, verapamil, quinidine, hydroquinidine, dispyramide, amiodarone, dofetilide, ibutilide, sotalol, pimazide, bepridil, cisapride, diphemanil, erythromycin, halofantrine, pentamidine, sparfloxacin, vincamine, alfuzosin, prazosin, terazosin, tamsulosin, amifostine
* Weight less than 45kg
* Pregnancy (Pre-menopausal women will only be entered into the study of they are surgically sterile or using effective birth control methods: These are abstinence for the period of the study, intrauterine contraception/device, male sexual partners with vasectomy)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2024-08-05 (Estimated); Study Completion 2024-08-05 (Estimated)

PRIMARY OUTCOMES:
Cognition as measured by the Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog) | 12 weeks
  The ADAS-Cog is used to determine the extent of cognitive decline in AD. It is a common cognitive testing instrument in clinical trials consisting of 11 tasks measuring disturbances in memory, language, praxis, attention and other cognitive abilities that are core symptoms of AD.

SECONDARY OUTCOMES:
Tests of Attention: Trails A and B | 12 weeks
  Neuropsychological test sensitive detecting cognitive impairment associated with dementia/AD.
Digit-symbol substitution | 12 weeks
  Neuropsychological test sensitive detecting cognitive impairment associated with dementia/AD.
Test of Everyday attention | 12 weeks
  Neuropsychological test sensitive detecting cognitive impairment associated with dementia/AD.
CANTAB-RVP | 12 weeks
  Neuropsychological test sensitive detecting cognitive impairment associated with dementia/AD.
Neuropsychiatric Inventory (NPI) | 12 weeks
  Examination and scoring of behavioural domains to determine the frequency and severity of behaviour with the patient and caregiver.
Zarit Burden Interview (22 Item) | 12 weeks
  Examination and scoring of behavioural domains to determine the frequency and severity of behaviour with the patient and caregiver.
Alzheimer's Disease Co-operative Study - Activities of Daily Living Inventory (ADCS-ADL) | 12 weeks
  Examination and scoring of behavioural domains to determine the frequency and severity of behaviour with the patient and caregiver.
Blood pressure | 12 weeks
  Measure of side effects.
Epworth Sleepiness Scale | 12 weeks
  Measure of side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Malhotra, MA BMBCh PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial Memory Unit, Charing Cross Hospital, London, United Kingdom

REFERENCES:
- [Derived] Hoang K, Watt H, Golemme M, Perry RJ, Ritchie C, Wilson D, Pickett J, Fox C, Howard R, Malhotra PA. Noradrenergic Add-on Therapy with Extended-Release Guanfacine in Alzheimer's Disease (NorAD): study protocol for a randomised clinical trial and COVID-19 amendments. Trials. 2022 Aug 1;23(1):623. doi: 10.1186/s13063-022-06190-3. PMID 35915506
- See also: HRA research summary — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/norad-version-10/